CLINICAL TRIAL: NCT06428448
Title: A Prospective, Multi-Center Study to Evaluate the Safety and Effectiveness of the REMEDY SPECTRUM IM Spacer Nail in the Treatment of Ankle-Related Infections
Brief Title: Study to Evaluate the REMEDY SPECTRUM IM Spacer Nail in the Treatment of Ankle-Related Infections
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OsteoRemedies, LLC (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-OR-001
Record Dates: First submitted 2024-05-17; First posted 2024-05-24 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Periprosthetic Joint Infection
Keywords: Ankle-related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects with REMEDY Spectrum IM Spacer Nail (Experimental): This is the REMEDY Spectrum IM Spacer Nail treatment group.
  Interventions: Combination Product: REMEDY Spectrum IM Spacer Nail

INTERVENTIONS:
Combination Product: REMEDY Spectrum IM Spacer Nail — The REMEDY SPECTRUM IM Spacer Nail is a single-use implant made of polymethylmethacrylate (PMMA) which is internally reinforced with a stainless-steel core (ASTM F138, ISO 5832-1). The PMMA of the REMEDY SPECTRUM IM Spacer Nail is laden with gentamicin and vancomycin.
  The nail has a slot at the distal end and can be combined with the surgeon's choice of fixation to prevent migration depending on the anatomy of the patient. The REMEDY SPECTRUM IM Spacer Nail is available in two lengths (150mm and 300mm) to accommodate variations in patient anatomy. The distal end has a threaded recess for mating with the optional distal cap, as well as the insertion and removal tools.

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of the REMEDY SPECTRUM IM Spacer Nail in the treatment of ankle-related infections. The study is expected to take approximately 18 months from first subject enrolled to the last follow-up visit. It will have a 12-month enrollment period and a 6-month follow-up. This study is a Prospective, multicenter, single-arm clinical trial. All subjects enrolled in this study will receive the REMEDY SPECTRUM IM Spacer Nail.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 21 years of age
2. Have an ankle-related infection
3. Is skeletally mature, as evidenced by closed epiphyses.
4. Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study
5. Be willing and able to comply with all study procedures including all pre-operative, post-operative requirements
6. If female and of child-bearing potential, must have a negative pregnancy test prior to the surgical procedure and no intention of becoming pregnant until study completion.

Exclusion Criteria:

1. Infections that do not involve the ankle
2. Have a known immunodeficiency; including subjects who are receiving or have received immunosuppressants, immunostimulating agents or radiation therapy within 6 months prior to surgery
3. Affected limb is dysvascular
4. Where adequate soft-tissue coverage cannot be achieved
5. Have any mental or psychological disorder that would impair their ability to complete the study questionnaires
6. Are currently pregnant or breastfeeding, or planning to become pregnant or breastfeed any time during the course of the study
7. Are currently a prisoner
8. Have any medical condition or other circumstances, in the judgment of the Investigator, that might interfere with the ability to return for follow-up visits, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the subject unable to perform appropriate post-operative activities.
9. History of vancomycin or gentamicin allergy
10. Are implanted with other antibiotic eluting products.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Successful Treatment of Infection Based on Lab Values and Culture | 6 months
  Healed wound and no infection recurrence caused by the same organism strain infection for duration of two weeks post antibiotic regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel McGuire Kennedy, Study Director — OsteoRemedies, LLC

IPD SHARING:
Plan to Share IPD: No